CLINICAL TRIAL: NCT00984022
Title: Aquacel vs. Iodoform Gauze for Filling Abscess Cavity Following Incision and Drainage: A Randomized Control Study
Brief Title: Aquacel Versus Iodoform Gauze for Filling Abscess Cavity Following Incision and Drainage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valleywise Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-003
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Abscess; Cellulitis
Keywords: abscess; MRSA; Aquacel dressing; Iodoform dressing
MeSH Terms: conditions — Abscess; Cellulitis

STUDY DESIGN:
Intervention Model Description: Aquacel vs. Iodoform Gauze
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodoform dressing (Active Comparator): Iodoform dressing for cutaneous abscess
  Interventions: Device: Type of dressing - Iodoform
- Aquacel dressing (Active Comparator): Aquacel dressing for cutaneous abscess
  Interventions: Device: Type of dressing - Aquacel

INTERVENTIONS:
Device: Type of dressing - Iodoform — Dressing for packing a cutaneous abscess
  Other Names: Iodoform
  Arms: Iodoform dressing
Device: Type of dressing - Aquacel — Aquacel dressing
  Other Names: Aquacel
  Arms: Aquacel dressing

SUMMARY:
This study compares Aquacel against routine Iodoform packing for packing abscess cavities after incision and drainage. It is hypothesized that Aquacel will produce speedier healing of the abscess.

DETAILED DESCRIPTION:
The large increase in the incidence of skin and soft tissue infections cause by methicillin resistant staphylococcus aureus (MRSA) has produced a corresponding increase in the number of ED patients presenting with abscesses that require incision and drainage. This study compares Aquacel against routine Iodoform packing for packing abscess cavities after incision and drainage. It is hypothesized that Aquacel will produce speedier healing of the abscess. More effective abscess healing will reduce the need for oral antibiotic coverage, which will in turn reduce the potential for drug resistance caused by indiscriminate use of oral antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* presenting to Maricopa Medical Center ED with cutaneous abscess requiring incision and drainage

Exclusion Criteria:

* known sensitivity to Aquacel
* pregnant, nursing, or expecting to become pregnant
* incarcerated patient
* prior treatment of same abscess with incision and drainage
* multiple abscesses
* immunodeficiency
* facial abscess
* suspected osteomyelitis or septic arthritis
* diabetic foot, decubitis, or ischaemic ulcers
* unable to provide informed consent or assent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2010-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Sinha, MD, Principal Investigator — District Medical Group
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Iodoform Dressing: Iodoform dressing for cutaneous abscess. Iodoform packing strips provided by Kendall, Curity, Tyco Healthcare Group LP, Mansfield, MA. Placed in the cavity after incision and drainage.
- Aquacel Dressing: Aquacel dressing for cutaneous abscess. Aquacel Ag ribbons (Conva Tec Ltd., Skillman, NJ). Placed in the cavity after incision and drainage.
Period: Overall Study
Arm/Group | Iodoform Dressing | Aquacel Dressing
Started | 43 | 49
Completed | 33 | 35
Not Completed | 10 | 14
Not completed — Lost to Follow-up | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iodoform Dressing | Aquacel Dressing | Total
Number analyzed (Participants) | 43 | 49 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 49 | 92
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (12.6) | 39.2 (11.6) | 38.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 28 | 33 | 61
Region of Enrollment [Number; unit: participants]
  United States | 43 | 49 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a 30% or Greater Reduction in Surface Area of Abscess
Description: Participants were assessed to see whether or not the surface area of the abscess was reduced by at least 30%, and the number of such participants is reported.
Time Frame: 2 weeks
Measure: Number; unit: Participants
Arm/Group | Iodoform Dressing | Aquacel Dressing
Number analyzed (Participants) | 43 | 49
Participants | 6 | 19
Statistical Analysis 1: Comparison: Iodoform Dressing vs Aquacel Dressing; The percentages achieving 30% or greater reduction in the surface area of the abscess were compared with Fisher's exact test; Test type: Superiority or Other; p = .0003, Fisher Exact

2. Secondary Outcome: Change in Patient Rating of Pain
Description: Change in mean pain score based on patient self-report, using Wong-Baker FACES pain rating scale. Scale ranges from 0 to 5, where 5 means the worst pain possible and 0 means no pain at all.
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Iodoform Dressing | Aquacel Dressing
Number analyzed (Participants) | 43 | 49
Scores on a scale | -1.23 (1.89) | -1.82 (1.73)
Statistical Analysis 1: Comparison: Iodoform Dressing vs Aquacel Dressing; Repeated measures ANOVA using 2 X 2 factorial design, with one between-subjects factor (Group) and one within-subjects factor (Time). Null hypothesis is: The type of dressing does not affect patient pain ratings; Test type: Superiority or Other; p = .043, ANOVA — Main effect for type of dressing

3. Secondary Outcome: Number of Participants Who Experienced a 30% or Greater Reduction in Surface Area of Cellulitis.
Description: Participants were assessed to see whether or not the surface area of the cellulitis was reduced by at least 30% and the number of such participants was reported.
Time Frame: 2 weeks
Measure: Number; unit: Participants
Arm/Group | Iodoform Dressing | Aquacel Dressing
Number analyzed (Participants) | 43 | 49
Participants | 13 | 13
Statistical Analysis 1: Comparison: Iodoform Dressing vs Aquacel Dressing; Fisher's exact test was used to compare the percentage of individuals achieving a 30% or greater reduction in cellulitis surface area between the Iodoform and Aquacel groups; Test type: Superiority or Other; p = .847, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Iodoform Dressing | Aquacel Dressing
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/49
Other Adverse Events (participants affected / at risk) | 0/43 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes